CLINICAL TRIAL: NCT04490382
Title: Evaluate Tactile Sensation and Proprioception in Lower Limb Amputees Using Neuromodulation
Brief Title: Spinal Cord Stimulation (SCS) for Amputees
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00102757
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Somatosensory Perception Following Lower Limb Amputation
Keywords: Neuromodulation; Phantom pain; Amputation
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients undergoing Neuromodulation (Experimental): Patients, who have had a lower limb amputation and undergoing neuromodulation as part of standard of care.
  Interventions: Device: 32 channel external stimulator

INTERVENTIONS:
Device: 32 channel external stimulator — Patients will be stimulated by the 32 channel external stimulator via leads placed as part of standard care neuromodulation. Then patients will undergo various tasks.

SUMMARY:
The purpose of this study is to investigate how leg amputee patients can feel sensations with neuromodulation while they are using a prosthetic leg. "Neuromodulation" is the process by which the nervous system can be regulated by targeted delivery of a stimulus, such as electrical stimulation or chemical agents, to specific neurological sites in the body. In this study, the investigators plan to use either electrical stimulation of the spinal cord (Spinal Cord Stimulation) or electrical stimulation of the dorsal root ganglion (DRG stimulation) as methods for neuromodulation.

Participation in this study will involve visiting the K-Lab (Human Performance Laboratory) at Duke's Sports Medicine Institute once prior to trial implant surgery, if feasible, and four times during the two weeks following the implantation of trial stimulation leads to evaluate sensations related to touch and position of the prosthetic leg as they are generated by neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject is able and willing to comply with the schedule and protocol
* Subject is a lower limb amputee who uses a prosthetic leg
* Subject is a good candidate for implantation of a stimulator for their amputation related pain
* Subject has stable neurological/cognitive function in the past 30 days
* Subject is able to provide informed consent

Exclusion Criteria:

* Subject is currently participating in a clinical investigation that includes an active treatment arm
* Subject currently has an active implantable device including an Implantable Cardioverter Defibrillator (ICD), pacemaker, spinal cord stimulator, or intrathecal drug pump
* Subject is a prisoner
* Female subject whom are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-20 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in stimulation as reported by patients | Visit 1(baseline), visit 2(up to six hours), visit 3(up to six hours), visit 4(up to six hours)
Change in stimulation parameters as measured by frequency | Visit 1(baseline), visit 2(up to six hours), visit 3(up to six hours), visit 4(up to six hours)
Change in stimulation parameters as measured by pulse width | Visit 1(baseline), visit 2(up to six hours), visit 3(up to six hours), visit 4(up to six hours)
Change in stimulation parameters as measured by amplitude | Visit 1(baseline), visit 2(up to six hours), visit 3(up to six hours), visit 4(up to six hours)
Change in pain score as measured by McGill Pain Questionnaire | Visit 1(baseline), visit 2(up to six hours), visit 3(up to six hours), visit 4(up to six hours)

SECONDARY OUTCOMES:
Change in gait parameters as measured by step frequency | Visit 1(baseline), visit 2(up to six hours), visit 3(up to six hours), visit 4(up to six hours)
Change in passive movement detection as measured by external sensors | Visit 1(baseline), visit 2(up to six hours), visit 3(up to six hours), visit 4(up to six hours)
Change in cortical reorganization measured by Electroencephalogram (EEG) | Visit 1(baseline), visit 2(up to six hours), visit 3(up to six hours), visit 4(up to six hours)

CONTACTS AND LOCATIONS:
Overall Officials: Nandan Lad, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No